CLINICAL TRIAL: NCT05193942
Title: Type 1 Hybrid Trial of Our Plan - a Brief, Couples-based HIV/STI Prevention Intervention
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Florida International University (Other)
Collaborators: University of Michigan (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: 3U54MD012393-05S2 (NIH)
Record Dates: First submitted 2021-11-17; First posted 2022-01-18 (Actual); Last update posted 2024-09-26 (Actual); Status verified 2024-09

CONDITIONS: HIV/AIDS
MeSH Terms: conditions — Acquired Immunodeficiency Syndrome

STUDY DESIGN:
Intervention Model Description: 4-month randomized controlled trial with an informational control condition
Who Masked: Participant
Masking Description: Participants (and their relationship partner) will not know in advance which arm (intervention, control) assigned to in the trial from randomization.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Intervention (Experimental): From baseline to 4-month post-test, participants in the intervention arm will have access to the Our Plan web app program.
  Interventions: Behavioral: Intervention Our Plan
- Informational control (Other): From baseline to 4-month post-test, participants in the informational control arm will not have access to the Our Plan web app program. Participants will instead receive a webpage with information about HIV/STI prevention options and resources to represent the current equivalent of a standard of care for online HIV resources.
  Interventions: Behavioral: Internation Informational Control

INTERVENTIONS:
Behavioral: Intervention Our Plan — From day 1 to day 120 (i.e., entire 4 month duration) of the trial, participants randomized to the intervention arm will be granted access and instructed to use the Our Plan program as directed. The Our Plan program includes modules covering topics of communication, decision-making, HIV/STI prevention, and stigma and discrimination. Each module contains content, questions, and activities for the participant and couple to complete. One goal of OurPlan is to help both partners of the couple create and use a risk- reduction plan of evidence-based prevention strategies over time. Answers provided during the assessments will help determine whether participants/couples created a risk-reduction plan and used evidence-based strategies over time, including changes in their own confidence, intention, and perceived ability to use these strategies.
  Arms: Intervention
Behavioral: Internation Informational Control — From day 1 to day 120 (i.e., entire 4 month duration) of the trial, participants randomized to the informational control condition will receive a webpage that contains information about HIV/STI prevention options and resources. This control condition represents the current equivalent of a standard of care for online HIV resources.
  Arms: Informational control

SUMMARY:
This webapp, couples-based HIV/STI prevention intervention project will use a Type 1 Hybrid Design Trial to determine efficacy to reduce HIV risk via uptake of evidence-based strategies and a tailored prevention plan among male couples who are in a new relationship (defined as 1 year or less). In addition, the project will be one of the first studies to investigate how intervention usage is associated with the outcomes over time, as well as explore best practices for future implementation and dissemination of such interventions by considering a variety of potential contexts. As such, the project is innovative, timely, and rigorous with sound scientific premise for helping to advance and bridge webapp HIV prevention science with existing community-level services.

DETAILED DESCRIPTION:
The beginning of a relationship (i.e., within first year) is a crucial time for male couples to make decisions about their HIV/STI and sexual health needs. Via a recently completed nation-wide pilot RCT, the theoretically-grounded, couples-based app intervention showed high acceptability and feasibility, and strong promise for encouraging 42 male couples to create a tailored, prevention plan consisting of evidence-based strategies that aligned with the dyad's HIV serostatus. Retention was 86%, signifying that both partners of each couple completed all assessments, used the app intervention as designed, and participated in an individual-level exit interview. Acceptability was >95%, and confirmed by using three different data sources (quantitative follow-up assessment, paradata from app intervention use, qualitative interview). The app intervention contained 4 modules (M1-M4) and a geo-locator sexual health resource finder. Although relationship partners individually used the app intervention (on their respective smartphones), questions and activities were built in each module to highlight within-couple comparisons and also encouraged couples to participate in discussion activities together. M1 was about enhancing communication and decision-making skills, while M2 focused on prevention strategies including creating a tailored prevention plan. M3 highlighted statistics of the HIV/STI epidemic, and M4 was about stigma and discrimination. Regarding promise, a two-fold increase was observed in the proportion of couples who created a tailored prevention plan when comparing baseline to follow-up assessment data, and while also considering their paradata. The next steps in this line of work would aim to improve the app intervention by integrating some of the acceptability feedback received, such as offering it in English and Spanish and adding content about importance of ART/PrEP adherence. Next steps also include, investigating - via mixed methods - how best to integrate the app intervention with local AIDS-service organizations (ASOs) and Community-based organizations (CBOs) for future scale up and improve use and adherence of evidence-based strategies among sexual minority men. Last but not least, a 4-month, Type 1 Hybrid Trial will be conducted to establish efficacy on couples' creation of a prevention plan, as well as participants' uptake of new evidence-based strategies (e.g., daily PrEP, regular testing, daily ART) and improving adherence of strategies currently in use. Findings from the Type 1 Hybrid Trial would inform best practices for integrating mHealth intervention science with brick-and-mortar services by including perspectives from the target population and ASOs/CBOs. The Type 1 Hybrid Trial study would occur in locations identified in Ending the HIV Epidemic Plan, such as Miami-Dade and Broward Counties in Florida.

ELIGIBILITY:
Inclusion Criteria:

* self-reported that currently self-identifies as a male
* self-reported in a sexual relationship with another self-identified male
* self-reported relationship length between 1 and 12 months
* self-reported anal sex with relationship partner in past month
* owns and uses an Internet-connected device (smartphone, tablet, computer)
* resides in the U.S.
* self-reported ability to read and understand English-language

Exclusion Criteria:

* Does not meet one or more of the inclusion criteria

Min Age: 18 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Gender Based: Yes — Cisgender men
Enrollment: 216 (Actual)
Dates: Start 2022-02-17 (Actual); Primary Completion 2023-09-30 (Actual); Study Completion 2023-09-30 (Actual)

PRIMARY OUTCOMES:
Change in creation of a detailed risk-reduction plan by comparing baseline response to month 4 response | Baseline, month 4
  At both time points, participants will be asked if they created a detailed risk-reduction plan that contains evidence-based strategies with their partner. Dichotomous measure: yes/no
Change in number of evidence-based prevention strategies being used over time by comparing baseline response to month 4 response | Baseline, month 4
  Participants will be asked how many evidence-based HIV/STI prevention strategies they are currently using at both time points.
Change in confidence about using evidence-based prevention strategies over time by comparing baseline response to month 4 response | Baseline, month 4
  Participants will be asked about their perceived confidence in using evidence-based HIV/STI prevention strategies at both time points. Validated theoretical measure (single item) with Likert-type scale response range of 1-5.
Change in intention to use evidence-based prevention strategies over time by comparing baseline response to month 4 response | Baseline, month 4
  Participants will be asked about their perceived intention to use evidence-based prevention strategies at both time points. Validated theoretical measure (single item) with Likert-type scale response range of 1-5.
Change in self-efficacy to use evidence-based prevention strategies over time by comparing baseline response to month 4 response | Baseline, month 4
  Participants will be asked about their perceived ability to use evidence-based prevention strategies at both time points. Validated theoretical measure (single item) with Likert-type response range of 1-5.

SECONDARY OUTCOMES:
Change in goal congruence on sexual health by comparing baseline response to month 4 response | Baseline, month 4
  Participants will be asked about their goal congruence regarding sexual health and their relationship partner at both time points. Validated theoretical measure containing 5 items, each containing a Likert-type response range of 1-5.
Change in mutual constructive communication by comparing baseline response to month 4 response | Baseline, month 4
  Participants will be asked about their mutual constructive communication patterns at both time points. Validated theoretical measure containing 3 items, each containing a Likert-type response range of 1-9.

CONTACTS AND LOCATIONS:
Locations (1):
- Florida International University, Miami, Florida, United States

IPD SHARING:
Plan to Share IPD: Yes
All IPD that underlie results in a publication
Supporting Information: Study Protocol, ICF, CSR
Time Frame: Starting 6 months after publication
Access Criteria: Interested research must email the PI with a request to access de-identified, anonymous IPD. The PI will review such requests for secondary analyses using de-identified data that have already been published.